CLINICAL TRIAL: NCT03741855
Title: Evaluating the Cloud DX Platform as a Tool for Self-management and Asynchronous Remote-monitoring of Chronic Obstructive Pulmonary Disease
Brief Title: Evaluating the Cloud DX Platform as a Tool for Self-management and Asynchronous Remote-monitoring of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Markham Stouffville Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WCHCDX-001
Record Dates: First submitted 2018-10-04; First posted 2018-11-15 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Self-Management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote-Monitoring Program (Experimental): Cloud Dx kit with remote-monitoring
  Interventions: Device: Cloud Dx Kit with remote-monitoring
- Self-Monitoring Program (Experimental): Cloud Dx kit with self-monitoring
  Interventions: Device: Cloud Dx Kit with self-monitoring
- Standard of Care (No Intervention): Participants will not be provided with the Cloud DX kit or an action plan

INTERVENTIONS:
Device: Cloud Dx Kit with self-monitoring — Patients in this group will be recording their vitals and symptoms with the Cloud DX platform everyday and will be provided with an action-plan that instructs them on what to do in response to their readings.
  Arms: Self-Monitoring Program
Device: Cloud Dx Kit with remote-monitoring — * Patients in this group will be recording their vitals and symptoms with the Cloud DX platform everyday and will be provided with an action-plan that instructs them on what to do in response to their readings.
  * A respiratory therapist (RT) will be monitoring asynchronously patient vitals and contacting them when their vitals exceed pre-determined thresholds.
  * The RT will also check on patients once a week irrespective of the value of the vitals.
  Arms: Remote-Monitoring Program

SUMMARY:
This study is an open-label, prospective, single-centre, randomized controlled trial, containing both a quantitative and a qualitative component and using a mixed-methods design. The study evaluates the impact of Cloud Dx kit, a device that can allows patients to monitor and manage Chronic Obstructive Pulmonary Disease (COPD) at their home. The study evaluates whether using Cloud Dx improves patients' COPD symptoms, ability to manage COPD, and quality of life.

It is anticipated that there will be 123 participants enrolled in this study across two experimental arms and one control arm. Participants will be in the study for 6 months and the study will run for 1 year a Markham-Stouffville Hospital. The primary outcome is the participants' self-management and activation which will be measured using The Partners in Health (PIH) scale, a validated scale measuring the current status of self-management, with items on knowledge of the condition and skills to monitor and respond to symptoms.

DETAILED DESCRIPTION:
This study is an open-label, prospective, single-centre, randomized controlled trial, containing both a quantitative and a qualitative component and using a mixed-methods design. The study evaluates the impact of Cloud Dx kit, a device that can allows patients to monitor and manage Chronic Obstructive Pulmonary Disease (COPD) at their home. The study evaluates whether using Cloud Dx improves patients' COPD symptoms, ability to manage COPD, and quality of life.

COPD is a pervasive disease that is estimated to affect 2.6 million Canadians (17%) aged 35 to 79 costing the healthcare system in Canada $1.5 billion annually. Ontarians living with COPD are frequent users of the health care system and account for 24% of hospital admissions and 24% of emergency department (ED) visits. COPD is responsible for the highest percentage (18.8%) of 30-day re-admissions to ED in the province.

A recent Cochrane review and meta-analysis concluded that remote monitoring has shown promise in reducing acute care utilization and reducing the number of exacerbations in COPD patients. While many studies have examined the effects of remote-monitoring, few studies have looked at how self-monitoring without clinical oversight affects patients' self-management skills and quality of life. Our goal is to compare a group of patients that are in both self- and remote-monitoring to a group of patients that are only in a self-monitoring program and compare each relative to a standard care group.

The technology used in this study is the Cloud Dx Connect Health Kit which will be used as a tool for self-monitoring and asynchronous remote-monitoring. It consists of a custom Tablet computer, Pulsewave® wrist cuff monitor, Oximeter, Scale and Therometer. Participants will use the kit to record daily their physiological and symptom readings.

This study will take place at Markham-Stoufville hospital with most patients being recruited from the Outpatient COPD Clinic (Respiratory Health-COPD Clinic) and will include patients who have a clinical diagnosis of COPD that has been diagnosed by their respirologist as per clinical guidelines. Recruitment will be ongoing until 123 patients have been recruited for the intervention phase. Once enrolled, participants will be randomized into one of three arms:

1. Self-Management group: Participants in this group will receive the Cloud Dx kit at the start of the study and will continue using it for 6 months. They will be recording their vitals and symptoms with the Cloud DX platform everyday and will be provided with an action-plan that instructs them on what to do in response to their readings.
2. Remote-Monitoring group: Participants in this group will receive the Cloud Dx kit at the start of the study and will continue using it for 6 months. They will be recording their vitals and symptoms with the Cloud DX platform everyday and will be provided with an action-plan that instructs them on what to do in response to their readings. In addition, a respiratory therapist (RT) will be monitoring asynchronously their vitals and contacting them when their vitals exceed pre-determined thresholds. The RT will also check on patients once a week irrespective of the value of the vitals.
3. Standard of care group: Participants will not be provided with a technology or an action plan (as the action plan is based on vitals and symptoms).

Primary and secondary outcomes will be assessed through a series of questionnaires at 3 time-points by all participants: at baseline, 3 months and 6 months.In addition, participants will also complete a demographic questionnaire at the initial visit.

Participants who expressed interest in the qualitative component will be invited to complete a qualitative interview. This qualitative process evaluation will occur alongside the quantitative component and will include 5 participants from the remote-monitoring group and 5 participants from the self-monitoring group. Healthcare providers involved in the care of participants will also be approached for participation in this evaluation process as well as upon study completion and will ideally include a sample of up to 5 providers and up to 5 hospital administrators and clinic managers

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD

Exclusion Criteria:

* Diagnosis of other significant lung disease (eg. interstitial lung disease) or dementia
* Lack of WiFi at home
* Inability to speak English
* Inability to use this technology due to physical or cognitive impairment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Self-management and Activation | 6 Months
  Measured with the Partners in Health Scale (PIHS)

SECONDARY OUTCOMES:
Quality of Life and Respiratory symptoms | 6 Months
  Assessed with the St. George's Respiratory Questionnaire (SGRQ)
Patient Knowledge of COPD | 6 Months
  Measured using the Bristol COPD Knowledge Questionnaire
COPD Assessment | 6 Months
  Measured by the COPD Assessment Test
Breathlessness | 6 Months
  Measured by the MRC Breathlessness Scale
Total number of contacts/calls to the outpatient clinic and deaths | 6 Months
  Recorded by RT; deaths caregiver reported
Total number of ED presentations, admissions to a hospital, exacerbations, visits to family doctor, number of nurse contacts, self-reported use of medication, self-reported smoking cessation | 6 Months
  self-reported
Total length of stay for all admissions (in days) | 6 Months
  self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Sacha Bhatia, Principal Investigator — Women's College Hospital
Locations (1):
- Markham-Stouffville Hospital, Markham, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in an academic peer-reviewed journal.
Supporting Information: Study Protocol, SAP
Time Frame: Link to protocol paper provided.
Access Criteria: Link to protocol paper provided.

REFERENCES:
- [Background] Evans J, Chen Y, Camp PG, Bowie DM, McRae L. Estimating the prevalence of COPD in Canada: Reported diagnosis versus measured airflow obstruction. Health Rep. 2014 Mar;25(3):3-11. PMID 24648134
- [Background] Gershon AS, Guan J, Victor JC, Goldstein R, To T. Quantifying health services use for chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2013 Mar 15;187(6):596-601. doi: 10.1164/rccm.201211-2044OC. Epub 2013 Jan 17. PMID 23328526
- [Background] Government of Canada, S. C. (2017, August 29). CANSIM - 105-0501 - Health indicator profile, annual estimates, by age group and sex, Canada, provinces, territories, health regions (2013 boundaries) and peer groups. Retrieved October 24, 2017, from http://www5.statcan.gc.ca/cansim/a26?lang=eng&id=1050501.
- [Background] McLean S, Nurmatov U, Liu JL, Pagliari C, Car J, Sheikh A. Telehealthcare for chronic obstructive pulmonary disease: Cochrane Review and meta-analysis. Br J Gen Pract. 2012 Nov;62(604):e739-49. doi: 10.3399/bjgp12X658269. PMID 23211177
- [Background] Mittmann N, Kuramoto L, Seung SJ, Haddon JM, Bradley-Kennedy C, Fitzgerald JM. The cost of moderate and severe COPD exacerbations to the Canadian healthcare system. Respir Med. 2008 Mar;102(3):413-21. doi: 10.1016/j.rmed.2007.10.010. Epub 2007 Dec 20. PMID 18086519
- [Derived] Stamenova V, Liang K, Yang R, Engel K, van Lieshout F, Lalingo E, Cheung A, Erwood A, Radina M, Greenwald A, Agarwal P, Sidhu A, Bhatia RS, Shaw J, Shafai R, Bhattacharyya O. Technology-Enabled Self-Management of Chronic Obstructive Pulmonary Disease With or Without Asynchronous Remote Monitoring: Randomized Controlled Trial. J Med Internet Res. 2020 Jul 30;22(7):e18598. doi: 10.2196/18598. PMID 32729843
- [Derived] Stamenova V, Yang R, Engel K, Liang K, van Lieshout F, Lalingo E, Cheung A, Erwood A, Radina M, Greenwald A, Agarwal P, Sidhu A, Bhatia RS, Shaw J, Shafai R, Bhattacharyya O. Technology-Enabled Self-Monitoring of Chronic Obstructive Pulmonary Disease With or Without Asynchronous Remote Monitoring: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Aug 19;8(8):e13920. doi: 10.2196/13920. PMID 31429418